CLINICAL TRIAL: NCT03504865
Title: Single-Blinded, Randomized Assessment of Post-Mastectomy Analgesia Using Exparel (Liposomal) Versus Standard Bupivacaine or Placebo
Brief Title: Post-Mastectomy Analgesia Using Exparel (Liposomal) Versus Standard Bupivacaine or Placebo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0175
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Mastectomy; Breast Cancer
Keywords: Exparel; Bupivacaine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Liposomal bupivacaine (Experimental): If a patient is randomized to the LB arm, at the appropriate time, under a surgeon's direction, 266 mg of (liposomal bupivacaine) LB in 20 cc of solution was expanded with various amounts of normal saline to cover the appropriate surgical field. Our routine expansion for a bilateral mastectomy is to add 80 mL of saline to 20 mL (266 mg) of LB. In our practice,we use an 18-gauge needle to inject the medication in a "field-effect" encompassing all 4 quadrants of the chest muscles (pectoralis and serratus) followed by injecting around the edges of the skin incision and drain site. This occurs prior to dissection of the pectoralis muscle and implant or tissue expander placement.
  Interventions: Drug: Liposomal bupivacaine
- Standard bupivacaine (Active Comparator): Patients randomized to the SB arm will receive weight-based dosing of bupivacaine, administered in the same manner as the LB arm.
  Interventions: Drug: Standard bupivacaine
- Placebo (Placebo Comparator): Patients who are in the placebo arm will have a similar volume of saline injected into the operative site.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Liposomal bupivacaine — Given at the end of the operation.
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: Standard bupivacaine — Given at the end of the operation.
  Arms: Standard bupivacaine
Other: Placebo — Saline will be administered as the placebo and will be given at the end of the operation.
  Arms: Placebo

SUMMARY:
This is a randomized, single-blinded placebo-controlled trial.

Patients will be randomized to one of three arms: (1) injection of liposomal bupivacaine at the end of the operation, (2) injection of standard bupivacaine at the end of the operation, or (3) no injection of local anesthetic. All patients will be able to receive IV and oral narcotic medications in the postoperative period on an as-needed basis.

If a patient is randomized to the LB arm, at the appropriate time, under a surgeon's direction, 266 mg of (liposomal bupivacaine) LB in 20 cc of solution was expanded with various amounts of normal saline to cover the appropriate surgical field. Our routine expansion for a bilateral mastectomy is to add 80 mL of saline to 20 mL (266 mg) of LB. In our practice,we use an 18-gauge needle to inject the medication in a "field-effect" encompassing all 4 quadrants of the chest muscles (pectoralis and serratus) followed by injecting around the edges of the skin incision and drain site. This occurs prior to dissection of the pectoralis muscle and implant or tissue expander placement.

Patients randomized to the SB arm will receive weight-based dosing of bupivacaine, administered in the same manner as the LB arm.

Patients who are in the placebo arm will have a similar volume of saline injected into the operative site.

Postoperatively, all patients will be kept in the hospital for at least one night. Total length of stay will be documented. They will all have the option of receiving IV morphine injections as well as oral acetaminophen-hydrocodone as needed for additional pain control. The administration of these additional medications will be recorded for each patient.

On postoperative day 1, each patient will be administered the American Pain Society Outcome Questionnaire while in the hospital. After discharge from the hospital, we will call the patient on postoperative day 2, 3, 5 and 7 to assess pain and satisfaction scores, using the same questions each time. For any patients staying in the hospital longer than 1 day, the questionnaire will be administered in the hospital on the same postoperative days. Subject participation only lasts for these 7 days of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. All female patients over 18
2. Subjects must be scheduled to undergo bilateral therapeutic or prophylactic skin or nipple-sparing mastectomy at Medstar Georgetown University Hospital
3. Subjects must have immediate reconstruction consisting of either tissue expander placement or direct implant placement at the time of mastectomy
4. subjects are capable of giving informed consent

Exclusion Criteria:

1. Subjects cannot be homeless persons
2. Subjects cannot have active drug/alcohol dependence or abuse history.
3. Subjects cannot be pregnant
4. Subjects cannot have documented chronic or recent opioid use as well as chronic pain syndromes
5. We will exclude any patients who will plan to undergo postoperative whole breast radiation
6. Subjects cannot have bupivacaine (and all related analog) allergies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Postop pain and satisfaction scores | 1 week
  Using a validated questionnaire - the American Pain Society Outcome Questionnaire
The Number of adverse events | 1 week
  As measured by number by the CTCAE v4.03

SECONDARY OUTCOMES:
Overall narcotic use | 1 week
  The amount of narcotics required per patient
Time in recovery | 1 week
  Measured as the number of hours from surgery to recovery
Time from recovery to discharge | 1 week
  Measured as the number of days and hours that a patient is admitted to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Tousimis, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No